CLINICAL TRIAL: NCT01249222
Title: Pro-inflammatory Cytokines Profile and Mortality Rate of Critically Ill Septic Patients Following Plasma Therapeutic Exchange
Brief Title: Pro-inflammatory Cytokines Profile and Mortality Rate of Critically Ill Septic Patients Following Plasmapheresis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Pharmaceutical Science research center, PSRC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-230-402
Record Dates: First submitted 2010-11-22; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Plasmapheresis; Plasma Exchange

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional treatment (No Intervention)
  Interventions: Other: plasmapheresis
- Plasmapheresis (Experimental)
  Interventions: Procedure: plasmapheresis; Other: plasmapheresis

INTERVENTIONS:
Procedure: plasmapheresis — Plasmapheresis was done every 24-48 hours and continues up to five times. Blood samples were collected 30 minutes before and after each session of plasmapheresis to determine sequential changes in plasma levels of IL-1β, IL-6 and TNF-α. During each exchange session a volume of 25-30 ml/kg bodyweight of patient's plasma was exchanged with equal volume of 20% human albumin diluted with normal saline solution. Before and after plasmapheresis, prothrombin time, activated partial thromboplastin time (aPTT), platelet count and serum calcium level were checked. calcium gluconate 10% (10 ml) was administered even if patient had normal serum calcium in order to prevent hypocalcaemia due to administration of citrate. All drugs except for vasopressors were stopped during procedure.
  Other Names: plasma exchange
  Arms: Plasmapheresis
Other: plasmapheresis — plasmapheresis 5 times every 24-48 hours. the apheresis volume will be 30 ml/kg.
  Other Names: plasma exchange

SUMMARY:
Sepsis is one of the most prevalent and fatal diseases in intensive care units .unfortunately, therapeutic approach to sepsis has remained unchanged for many years. Nowadays, the role of cytokines in pathogenesis of sepsis is obvious. Continuous elevated levels of various cytokines in severe sepsis could result in uncontrolled inflammation status. Breaking of inflammatory cascade may lead to improvement in survival. It seems that modulation of inflammation is one of the strategic plans to conquest sepsis. Therefore, elimination of bacterial toxins and pro-inflammatory cytokines from the systemic circulation by plasmapheresis supposed to be rational approach.

Researchers have done several attempts to clarify the efficacy of plasmapheresis in sepsis treatment. However because of inconsistent results, routine use of this procedure in patients with severe sepsis remains controversial.

The aim of the present survey is to determine the effect of plasmapheresis on plasma levels of main pro-inflammatory cytokines and evaluate its therapeutic efficacy in improvement of outcome and treatment of severe sepsis.

DETAILED DESCRIPTION:
Method 27 patients with sepsis less than 24 hours, admitted in ICU, 16- 60 years old, male and female, randomized divided two groups(P=12, S=15) study in randomized clinical trial.

Inclusion criteria:

A: At least 3 of SIRS criteria;

1. 36> Tem> 38 ◦c
2. HR>90 bpm (without medication)
3. RR>20 bpm or PaCo2≤ 32 on mechanical ventilation
4. WBC<4000 or >12000 or > 10% immature neutrophil

B: Documented diagnosis of sepsis (separation organism from blood, urine, CSF, secretions such as trachea and sore) or strong suspect for infection with at least one of following:

1. WBC in sterile area,
2. Perforated viscera,
3. Radiological evidences of pneumonia,
4. High risk of infection such as cholangitis. Severity of disease is appointed with APACHE II (on result of laboratories in last 24 hours)

Exclusion criteria:

1. Pass more than 24 hours from diagnosis of sepsis.
2. High likelihood of mortality (renal failure, hepatic encephalopathy, ….) or imminent death(APACHE II score >25)
3. Pregnant or lactescent woman
4. 16 > age years old
5. No satisfaction of patient

Treatments of S group include:

1. Early goal - directed resuscitation
2. Appropriate diagnostic studies prior to antibiotics
3. Early broad - spectrum antibiotics
4. Narrowing antibiotic therapy based on microbial therapy and clinical data
5. Source control
6. Stress dose steroids for septic shock
7. Target Hb values of 7-9 g/dl in absence of coronary artery disease or acute hemorrhage
8. Lung protective ventilation for ALI/ARDS
9. Avoidance of Neuromuscular blockade
10. Maintenance of blood glucose < 150mg/dl
11. DVT/stress ulcer prophylaxis

In plasmapheresis (P) group, plasmapheresis will add into conventional therapy which is mentioned above. volume of plasmapheresis is 20-40 ml/Kg with five time in a week (distance 24-48 hours) that will do with speed of 60-120 ml/min through of central venous catheter.

Steps of plasmapheresis:

1. calculation of plasma volume
2. PT, PTT, Plt before and after plasmapheresis
3. Replacement plasma with albumin 20% and/or normal saline
4. Check of serum calcium before and after plasmapheresis. Injection of calcium gluconate 10%.
5. Stop of all of drugs (except vasopressor)
6. Cardiovascular monitoring during plasmapheresis
7. Infusion of heparin 500 u/h Demographic characters of patients (age, sex, weight, BMI) will record. Central venous, arterial line and Foley catheter will insert. For all of patients will do follow assays daily: CVP, BP, ABG, BUN, Cr, Na, K, CBC, PLT, PT, PTT, U/A, P, Ca, Mg, Chest X Ray. LFT and Alb

Level of biomarkers evaluate at 1st, 3rd, 5th, 7th and 14th day of study. In P group, evaluation will do before and after of plasmapheresis. Biomarkers include:

1. TNF-α (early release cytokine)(plasma)
2. IL-1 (early release cytokine)(plasma)
3. IL-6 (pro & anti-inflammatory cytokine)(plasma) Patient will evaluate for 14 days or until death. Patient's morbidity will record until 30 days.

Evaluation of morbidity will do by scoring systems:

* TISS score (Therapeutic intervention scoring system): for evaluation of severity of care.
* SOFA score (Sepsis- related organ function assessment): for evaluation of organ function.
* ADL score (Activities of daily living) Recorded information will analyze by t- test for quantitative variables and χ 2 square for qualitative variables, with α = 0/05.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis criteria which were defined by the ACCP/SCCM consensus conference

Exclusion Criteria:

* Post CPR, pregnant and under 16 years old patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mojtaba Mojtahedzadeh, Ph.D, Study Chair — 1Department of Clinical Pharmacy, Faculty of Pharmacy and Pharmaceutical Sciences Research Center, Tehran University of Medical Sciences, Tehran, Iran.
Locations (1):
- Tehran University of Medical sciences, Imam hospital, Tehran, Tehran Province, Iran